CLINICAL TRIAL: NCT04344691
Title: Relation Between Rectus Femoris Muscle Tension and Hamstring Strength and Activity in Healthy Sprinters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Pablo Fanlo, Principal Investigator, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-001
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Muscle Stretching Exercise
Keywords: muscle length; strength; sprint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 5 minutes waiting time
- Stretching (Experimental): Rectus femoris static stretching during 90' (with three hold-relax progressions until final ROM)
  Interventions: Procedure: Rectus femoris stretching

INTERVENTIONS:
Procedure: Rectus femoris stretching — Patient lying prone with the non-implicated leg outside the treatment table resting on the floor. Physical therapist flexes patients knee until tension is felt. In that position 5 seconds' isometric contraction is asked and physical therapist progresses in knee flexion range of motion until new tension is felt. After three contract-relax procedures physical therapist holds the range of motion for 30 seconds.
  Arms: Stretching

SUMMARY:
An open-label, single-group, control, pretest-posttest clinical trial is going to be conducted, with 16 healthy sprinters. Rectus femoris length and hamstring strength and electromyography is going to be assessed at baseline, after 10 minutes control and after an static rectus femoris stretching technique.

The main objective is to register if an increase in rectus femoris stretching Range of Motion, increases hamstring strength and activity due to their antagonic relationship and their relation with pelvic tilt.

ELIGIBILITY:
Inclusion criteria:

* The athletes recruited have to be under regular training and competition
* Free of any symptoms, at least 3 days training weekly for the last three years
* Give written consent

Exclusion criteria:

- Subjects who have suffered lower limb or back injuries during those last three years

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Rectus femoris length | Inmediate after intervention; up to 10 minutes
  Knee flexion range of motion with inclinometer
Biceps femoris strength | Inmediate after intervention; up to 10 minutes
  Dynamometry
Gluteus maximus strength | Inmediate after intervention; up to 10 minutes
  Dynamometry

SECONDARY OUTCOMES:
Rectus femoris tensomyography | Inmediate after intervention; up to 10 minutes
  tensomyography
Pelvic anteversion | Inmediate after intervention; up to 10 minutes
  Photometry of lateral view
Sprint muscle activity | Inmediate after intervention; up to 10 minutes
  Electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Alazne Ruiz de Escudero Zapico, PhD, Principal Investigator — Universidad Pública de Navarra
Locations (1):
- Cnetro ragonés del Deporte, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Principal investigator will review requests and criteria for reviewing requests will be individually assessed